CLINICAL TRIAL: NCT02158390
Title: Phenotypic Specific Communication Intervention for Children With Down Syndrome
Acronym: Merck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Ann Kaiser, Susan W. Gray Professor of Education and Human Development, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05302014
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Language Impairment; Down Syndrome
Keywords: Down syndrome; Language intervention; Communication intervention
MeSH Terms: conditions — Language Disorders; Down Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Jasper-EMT with words and AAC (Experimental): Jasper-EMT with words and AAC
  A therapist plus parent implemented social communication intervention which include use of the iPad for a mode of communication. A total of 6 hour long workshops with the parent and 42 hour long intervention sessions with the child occur; half include the parent as therapist and occur in the home. The treatment lasts approximately 4 months.
  Interventions: Behavioral: Jasper-EMT with words and AAC
- Community treatment as usual (No Intervention): Children access educational and speech-language interventions available to them through schools and community resources.

INTERVENTIONS:
Behavioral: Jasper-EMT with words and AAC — Jasper-EMT with words and AAC
  A therapist plus parent implemented social communication intervention which include use of the iPad for a mode of communication. A total of 6 hour long workshops with the parent and 42 hour long intervention sessions with the child occur; half include the parent as therapist and occur in the home. The treatment lasts approximately 4 months.
  Arms: Jasper-EMT with words and AAC

SUMMARY:
Children with Down syndrome (DS) have greater difficulty acquiring expressive language than is predicted by their general cognitive abilities and language comprehension (Miller, 1999). To date, interventions to improve communication outcomes for children with DS have met with only modest success. The proposed study is a randomized controlled trial of an early communication intervention combining two evidence-based treatments that teach expressive communication (Enhanced Milieu Teaching; EMT) and joint attention/symbolic play (Joint Attention Symbolic Play Engagement and Regulation; JASPER) using a dual mode (words +AAC). The intervention (a) teaches the foundations of communication (joint attention, play), (b) builds on positive child characteristics of social attention, (c) uses naturalistic strategies to increase the rate and complexity of communication and increase task engagement, (d) addresses the potential value of adding visual support (AAC) to spoken communication, and (e) includes parents as implementers of the intervention to promote generalization across settings and activities, and to ensure maintenance over time. It is hypothesized that children with DS enrolled in the intervention will have better language and communication skills at the end of treatment and followup than children in the BAU comparison group.The study will enroll 82 30 to 54 month old children with DS who have fewer than 20 words. Examining predictors of response to treatment and the effects of treatment on executive functioning will inform both theory and practice.

DETAILED DESCRIPTION:
This is a two-site randomized controlled trial (RCT) of the efficacy of JASP-EMT, an innovative blended communication intervention, JASPER (joint engagement and play intervention), and EMT (Enhanced Milieu Teaching). The study evaluates the relative benefits of teaching young children with DS using dual communication modes: spoken words with AAC. JASP-EMT involves direct intervention with children as well as parent training in an attempt to increase generalization of intervention effects. A control group will receive community treatment as usual (BAU). Participants include 82 children with DS ages 30 to 54 months across two sites.

AIM 1: To examine the effects of an experimental intervention (Words + AAC) on primary (expressive language) and secondary outcomes (receptive language, symbolic play, symbol-infused joint engagement, and parent use of language support strategies).

H1: Children in the Words+AAC group will have significantly better primary and secondary outcomes than children in the control group.

H2: Parents of children in Words+AAC group will demonstrate increased use of language support strategies than parents of children in the control group.

AIM 2: To examine maintenance and generalization of the effects of the experimental interventions on children and their parents.

H3: Intervention effects will maintain at follow-up and generalize across contexts.

AIM 3 (exploratory): To examine the effect of potential child level moderators on the primary and secondary outcomes of the study.

H4: Child characteristics at baseline (e.g., speech intelligibility, cognitive level) will moderate primary child outcomes.

AIM 4 (exploratory): To examine the effect of the experimental intervention on executive functioning.

H5: Children in the Words+AAC group will demonstrate improved executive functioning following intervention relative to the children in the control group.

Participants

A total of 82 children and their parents will be recruited to the study (41 at Vanderbilt and 41 at UCLA). Child MA of 18 months ensures children have the cognitive skills for symbolic representation in communication. The sample is expected to be 40% minority with equal numbers of males and females. Most parents are expected to be lower to upper middle class mothers.

Summary of Intervention

The goal of the intervention is to help children with DS develop expressive language skills that will improve participation in social, academic and community environments. Children will receive direct intervention from a therapist; additionally, parents will be taught to use the Words + AAC strategies in the clinic and at home across routines. Therapists use all strategies throughout the intervention; parents learn strategies sequentially.

Length of Intervention: 4/week for 4 months (48 sessions); 40 minute clinic sessions, 60 minute home sessions Type of Intervention sessions: 6 workshops, 18 clinic training sessions, 24 home training sessions Mode: AAC (iPad) and verbal input and output Maintenance: every six weeks for 6 months after completion of the intervention

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of DS from medical records.
2. Mental age (MA) of 18 months as measured on the Visual Reception subtest of the Mullen Scales of Early Learning.
3. Expressive vocabulary of fewer than 20 words at measured on a naturalistic language sample.
4. Age between 30 and 54 months
5. English or Spanish as the primary language at home.
6. Parents who are willing to participate in parent training.

Exclusion Criteria:

1. Major medical conditions other than DS, specifically (a) developmental disorders (e.g. autism); (b) sensory disabilities (e.g. blindness/deafness), and (c) motor disabilities not related to DS, (e.g. cerebral palsy)

-

Ages: 30 Months to 54 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2014-06; Primary Completion 2017-08-30 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
Spoken language | up to 3 months
  Spoken language is measured by transcribing child utterances ( spoken and AAC generated ) during 20 minute naturalistic language samples. Linguistic analysis are automated, via SALT.

SECONDARY OUTCOMES:
Receptive language | up to 3 months
  Receptive language is assessed by child performance on the Preschool Language Scale 5th Edition ( PLS-5), a standardized language assessment.
Executive Functioning | up to 3 months
  Children's executive functioning abilities will be assessed across a variety of tasks measuring persistence, planning, and attention.

OTHER OUTCOMES:
Parent use of Joint Attention Symbolic Play Engagement and Regulation- Enhanced Milieu Teaching ( Jasper-EMT) strategies | up to 3 months
  Observations of parent-child interactions are coded to determine parent use of key intervention strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Ann P Kaiser, PhD, Principal Investigator — Vanderbilt University; Connie Kasari, PhD, Study Director — University of California, Los Angeles
Locations (2):
- United States (2):
  - University of California, Los Angeles Center for Autism Research and Treatment, Los Angeles, California
  - Vanderbilt University Kennedy Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
This project does not require a data sharing plan. Results will be reported on profession journals.